CLINICAL TRIAL: NCT02848183
Title: Optimal Treatment Strategy Based on Prognostic Groups for Pediatric de Novo Acute Myeloid Leukemia
Brief Title: Optimal Treatment Strategy Based on for Pediatric AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 2015-11-028
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Pediatric Acute Myeloid Leukemia
MeSH Terms: interventions — Cytarabine; Idarubicin; Mitoxantrone; Etoposide; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pediatric de novo acute myeloid leukemia (Experimental): I. Chemotherapy Induction-1: Cytarabine + idarubicin Induction-2: High dose (HD) cytarabine + mitoxantrone Consolidation-1: Cytarabine + idarubicin Consolidation-2: HD cytarabine + etoposide Consolidation-3: HD cytarabine + mitoxantrone Consolidation-4: HD cytarabine + etoposide
  II. Allogeneic hematopoietic stem cell transplantation (HSCT) Favorable prognosis group: chemotherapy only Intermediate prognosis group: chemotherapy or HSCT with reduced intensity conditioning Poor prognosis group: HSCT with myeloablative conditioning
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Mitoxantrone; Drug: Etoposide; Procedure: Hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: Cytarabine
Drug: Idarubicin
Drug: Mitoxantrone
Drug: Etoposide
Procedure: Hematopoietic stem cell transplantation

SUMMARY:
The purpose of this study is to optimize therapy according to the known risk factors and treatment response in pediatric acute myeloid leukemia (AML)

DETAILED DESCRIPTION:
I. Risk group assessment Favorable prognosis group: Low risk features + Good response

Intermediate prognosis group:

1. Low risk features + Delayed response-1
2. Standard risk features + Good response
3. Standard risk features + Delayed response-1

Poor prognosis group:

1. Any high risk features irrespective of treatment response
2. Any delayed response-2 irrespective of risk features
3. Any refractory state irrespective of risk features
4. Any early relapse

II. Chemotherapy Induction-1: Cytarabine + idarubicin Induction-2: High dose (HD) cytarabine + mitoxantrone Consolidation-1: Cytarabine + idarubicin Consolidation-2: HD cytarabine + etoposide Consolidation-3: HD cytarabine + mitoxantrone Consolidation-4: HD cytarabine + etoposide

III. Allogeneic hematopoietic stem cell transplantation (HSCT) Favorable prognosis group: chemotherapy only Intermediate prognosis group: chemotherapy or HSCT with reduced intensity conditioning Poor prognosis group: HSCT with myeloablative conditioning

ELIGIBILITY:
Inclusion Criteria:

* Patients who were newly diagnosed with de novo AML
* Patients who had recurrent cytogenetic abnormalities of AML even though the bone marrow blast percent is lower than 20%

Exclusion Criteria:

* Acute promyelocytic leukemia
* Down syndrome AML
* Therapy-related AML
* AML developed from myelodysplastic syndrome or other marrow failure syndrome
* Isolated myeloid sarcoma without bone marrow involvement
* Patients who cannot undergo chemotherapy as scheduled due to serious complications at diagnosis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Rate of event free survival | Up to 5 years

SECONDARY OUTCOMES:
Proportion of patients who achieved complete remission | Up to 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Chonnam National University Hwasun Hospital, Chonnam
  - Samsung Medical Center, Seoul
  - St. Mary Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No